CLINICAL TRIAL: NCT04275661
Title: Efficacy and Safety of Ketamine Versus Magnesium Sulphate as Adjuvants to Levobupivacaine in Ultrasound (US) Bi-level Erector Spinae Block in Breast Cancer Surgery
Brief Title: Ketamine Versus Magnesium Sulphate as Adjuvants for ESPB in Breast Cancer Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Rabiee Ali, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ESPB in breast cancer surgery
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Analgesia; Breast Cancer
MeSH Terms: conditions — Agnosia; Breast Neoplasms | interventions — High-Energy Shock Waves; Levobupivacaine; Ketamine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group (C) (control group) (Placebo Comparator): Patient will receive 10 ml 0.25% levobupivacaine into interfascial plane below erector spinae muscle at level of T5 and 10 ml at level of T7.
  Interventions: Procedure: Ultrasound (US) bi-level erector spinae block; Drug: levobupivacaine
- Group (K) (Ketamine group) (Experimental): Patient will receive 10 ml 0.25% levobupivacaine into interfascial plane below erector spinae muscle at level of T5 and 10 ml at level of T7+ 1 mg / kg ketamine at each level with total dose 2mg/kg
  Interventions: Procedure: Ultrasound (US) bi-level erector spinae block; Drug: levobupivacaine; Drug: Ketamine
- Group (M) (magnesium sulphate group) (Experimental): Patient will receive 10 ml 0.25% levobupivacaine into interfascial plane below erector spinae muscle at level of T5 and 10 ml at level of T7+ 1 mg / kg MgSo4 at each level with total dose 2mg/kg
  Interventions: Procedure: Ultrasound (US) bi-level erector spinae block; Drug: levobupivacaine; Drug: Magnesium Sulfate

INTERVENTIONS:
Procedure: Ultrasound (US) bi-level erector spinae block — nerve block
Drug: levobupivacaine — 20 ml 0.25% levobupivacaine injected into fascial plane deep to erector spinae muscle
Drug: Ketamine — 2 mg /kg ketamine.injected into fascial plane deep to erector spinae muscle
  Arms: Group (K) (Ketamine group)
Drug: Magnesium Sulfate — 2mg/kg Magnesium Sulfate .injected into fascial plane deep to erector spinae muscle
  Arms: Group (M) (magnesium sulphate group)

SUMMARY:
Our aim will be to compare the analgesic efficacy and safety of ketamine and magnesium sulphate as adjuvants to levobupivacaine in erector spinae plane block in modified radical mastectomy.

DETAILED DESCRIPTION:
The participating females will be randomly allocated using computer generated randomizer program (http://www.randomizer.org) into one of 3 groups.

Group (C) / (I): 20 patients (control group):

Patient will receive 20 ml 0.25% levobupivacaine into interfascial plane below erector spinae muscle at level of T5 and T7.

Group (K) / (II): 20 patients (Ketamine group):

Patient will receive 20ml 0.25% levobupivacaine as above + 2 mg /kg ketamine.

Group (M) / (III): 20 patients (magnesium sulphate group):

Patient will receive 20ml 0.25% levobupivacaine as above + 2mg/kg MgSo4.

Study protocol:

Premedication will be given, after complete fasting hours after applying standard monitors (noninvasive blood pressure, pulse oximetery. ECG, temp, and capnography), an intravenous cannula will be placed and secured in the opposite side to surgery.

Ultrasound guided Erector spinae plane (ESP) block will be given with patient in sitting position depending on surgical site (lt. or Rt.) ESP block will be given using high frequency linear u/s transducer, the probe is placed in longitudinal orientation lateral to thoracic fifth and seventh spinous process, then Trapezious m., Rhomboideus major muscle, and erector spinae muscle, are identified from surface, we will deposite 20 ml of 0.25% levobupivacairen into interfacial plane below erector spinae muscle.

General anesthesia will be induced with lμg/kg fentanyl, 2mg/kg propofol, 0.5 mg/kg atracurium inhalational anesthesia (isoflurane or sevoflurane)

1gm paracetamol after induction No other narcotic, analgesic or sedative will be administrated during operative period.

Standard monitor (MABP, HR , SaO2 & EtCo2) will be observed and recorded every 30 min till end of surgery Post-operative ; the patient will be transferred to the post anesthesia care unit (PACU). In PACU the following data included heart rate, mean blood pressure, respiratory rate and oxygen saturation and VAS scores (at rest and after movement in the form of abduction of ipsilateral arm ) at baseline,2,4,6,12,24 and 48 hours post-operatively to evaluate acute pain will be observed and recorded. The attending anesthesiologist, surgeon and the data collecting personal will be unaware of the patient assignment.

Rescue post-operative analgesia in the form of morphine Patient controlled analgesia (PCA ) with an initial bolus of 0.1 mg/ kg morphine once pain is expressed followed by 1mg bolus with a locked period of 15 minutes with no back ground infusion allowed. The time to first request of analgesia and the total analgesic consumption in the 1st 48 hour will be observed and recorded. Postoperative adverse effects will be observed and treated

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 60 years.
* ASA grade I - II.

Exclusion Criteria:

* Patient refusal. known allergy to the study drugs skin infection at site of needle puncture significant organ dysfunction Coagulopathy drug or alcohol abuse psychiatric illness that would interfere with perception and assessment of pain.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
total morphine consumption in first 48 hours | 48 hours
  determine the analgesic effect of ketamine and magnesium sulphate in decreasing morphine consumption
time to first request of analgesia | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: khaled fares, Study Director — Assiut University; hamdy abbas, Study Director — Assiut University; fatma adel, Study Director — Assiut University
Locations (1):
- south Egypt Cancer Institute Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Gumus Demirbilek S. Bi-level erector spinae plane block for the control of severe back pain related to vertebral metastasis. BMJ Case Rep. 2019 Jun 20;12(6):e228129. doi: 10.1136/bcr-2018-228129. PMID 31227568
- [Background] Kwon WJ, Bang SU, Sun WY. Erector Spinae Plane Block for Effective Analgesia after Total Mastectomy with Sentinel or Axillary Lymph Node Dissection: a Report of Three Cases. J Korean Med Sci. 2018 Nov 5;33(45):e291. doi: 10.3346/jkms.2018.33.e291. No abstract available. PMID 31044575
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005